CLINICAL TRIAL: NCT02849587
Title: A Randomized, Controlled Trial of Cannabis in Healthy Volunteers Evaluating Simulated Driving, Field Performance Tests and Cannabinoid Levels
Brief Title: The Impact and Detection of Driving Impairments Associated With Acute Cannabis Smoking
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Thomas D. Marcotte, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 160641
Record Dates: First submitted 2016-07-14; First posted 2016-07-29 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Cannabis Intoxication
Keywords: Driving Under the Influence; Memory Impairment; Reaction Time; Time Perception; Cannabis; Marijuana; Whole Blood; Oral Fluid; Breath; Driving simulator
MeSH Terms: conditions — Driving Under the Influence; Memory Disorders; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to smoke a cannabis cigarette containing placebo (.02%), 5.9% or 13.4% THC.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Product will be dispensed from the Research Pharmacy. All assessors, investigators, and participants are blinded to the THC content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Cannabis (Placebo Comparator): Subjects will smoke cannabis with placebo THC (.02%) ad libitum
  Interventions: Drug: Cannabis
- Cannabis with 5.9% THC (Experimental): Subjects will smoke cannabis cigarettes with 5.9% THC ad libitum
  Interventions: Drug: Cannabis
- Cannabis with 13.4% THC (Experimental): Subjects will smoke cannabis cigarettes with 13.4% THC ad libitum
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Participants will smoke a cannabis cigarette ad libitum as per their usual routine
  Other Names: Marijuana

SUMMARY:
This study was authorized by the California Legislature (Assembly Bill 266, the Medical Marijuana Regulation and Safety Act to help with detection of driving under the influence of cannabis. One hundred and eighty healthy volunteers will inhale smoked cannabis with either 0% (placebo), 5.9%, or 13.4% Δ9-tetrahydrocannabinol (THC) at the beginning of the day, and then complete driving simulations, iPad-based performance assessments, and bodily fluid draws (e.g., blood, saliva, breath) before the cannabis smoking and a number of times over the subsequent 6 hours after cannabis smoking. The purpose is to determine (1) the relationship of the dose of Δ9-THC on driving performance and (2) the duration of driving impairment in terms of hours from initial use, (3) if saliva or expired air can serve as a useful substitute for blood sampling of Δ9-THC, and (4) if testing using an iPad can serve as a useful adjunct to the standardized field sobriety test in identifying acute impairment from cannabis.

DETAILED DESCRIPTION:
There are several studies that suggest higher doses of whole-blood Δ9-tetrahydrocannabinol (Δ9-THC) concentration are associated with increased crash risk and crash culpability. However, attempts to define a cut-off point for blood Δ9-THC levels have proven to be challenging. Unlike alcohol, for which a level can be reasonably measured using a breathalyzer (and confirmed with a blood test), detection of a cut-off point for intoxication related to Δ9-THC concentration has eluded scientific verification. Recent evidence suggests blood Δ9-THC concentrations of 2-5 ng/mL are associated with substantial driving impairment, particularly in occasional smokers. Others have countered that this level leads to false positives, particularly in heavy cannabis users inasmuch as THC may be detectable in their blood specimens for 12-24 hours after inhalation. Given that 12 to 24 hours is beyond the likely period of driving impairment, this would appear to be a justifiable objection to a per se cut-off point for a Δ9-THC concentration indicative of impairment. Maximal driving impairment is found 20 to 40 minutes after smoking, and the risk of driving impairment decreases over the following hours, at least in those who smoke 18 mg Δ9-THC or less, the dose often used experimentally to duplicate a single joint. Other studies, however, report residual motor vehicle accident crash risk when cannabis is used within 4 hours prior to driving.

The roadside examination using the Standardized Field Sobriety Test (SFST) for proof of cannabis-related impairment has not been an ideal alternative to blood levels. Originally devised to evaluate impairment under the influence of alcohol, the SFST is comprised of three examinations administered in a standardized manner by law enforcement officers. The 'Horizontal Gaze Nystagmus' (HGN), the 'One Leg Stand' (OLS) and the 'Walk and Turn' test (WAT) require a person to follow instructions and perform motor activities. During the assessments, officers observe and record signs of impairment. In one study, Δ9-THC produced impairments on overall SFST performance in 50 % of the participants. In a separate study involving acute administration of cannabis, 30% of people failed the SFST. This discrepancy was thought to be in part due to the participant's cannabis use history, as well as low percentage of THC in the cannabis. The reported frequency of cannabis use varied from once a week to once every 2-6 months in the study where there was a failure on the SFST by 50% of the participants. The other study included more frequent users who smoked cannabis on at least four occasions per week.

Based upon the above, another means is needed to help law enforcement officers discern driving under the influence of cannabis. One future possibility is the development of performance-based measures of cannabis-related impairments. This will include testing of critical tracking, time estimation, balance and visual spatial learning. The investigators have selected brief measures in order to be practicably administered repeatedly over a short time period, as well as tests that have the potential to translate to a field-feasible tablet-based format, should there be benefit in possibly including these in future performance-based measures for use in the field by law enforcement officers (e.g., a cannabis-focused field sobriety test).

ELIGIBILITY:
Inclusion Criteria:

* Be a licensed driver.
* Need to have acuity of 20/40 or better, with or without correction on a Snellen Visual Acuity eye chart.

Exclusion Criteria:

* At the discretion of the examining physician, individuals with significant cardiovascular, hepatic or renal disease, uncontrolled hypertension, and chronic pulmonary disease (eg, asthma, COPD) will be excluded.
* Unwillingness to abstain from cannabis for 2 days prior to screening and experimental visits
* Positive pregnancy test
* A positive result on toxicity screening for cocaine, amphetamines, opiates, and phencyclidine (PCP) will exclude individuals from participation.
* Unwilling to refrain from driving or operating heavy machinery for four hours after consuming study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Marcotte, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Center for Medicinal Cannabis Research, UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to facilitate meta-analyses
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon manuscript publications
Access Criteria: Approved researchers

REFERENCES:
- [Background] Hartman RL, Huestis MA. Cannabis effects on driving skills. Clin Chem. 2013 Mar;59(3):478-92. doi: 10.1373/clinchem.2012.194381. Epub 2012 Dec 7. PMID 23220273
- [Background] Papafotiou K, Carter JD, Stough C. An evaluation of the sensitivity of the Standardised Field Sobriety Tests (SFSTs) to detect impairment due to marijuana intoxication. Psychopharmacology (Berl). 2005 Jun;180(1):107-14. doi: 10.1007/s00213-004-2119-9. Epub 2004 Dec 24. PMID 15619106
- [Background] Fabritius M, Chtioui H, Battistella G, Annoni JM, Dao K, Favrat B, Fornari E, Lauer E, Maeder P, Giroud C. Comparison of cannabinoid concentrations in oral fluid and whole blood between occasional and regular cannabis smokers prior to and after smoking a cannabis joint. Anal Bioanal Chem. 2013 Dec;405(30):9791-803. doi: 10.1007/s00216-013-7412-1. Epub 2013 Nov 8. PMID 24202191
- [Background] Beck O, Stephanson N, Sandqvist S, Franck J. Detection of drugs of abuse in exhaled breath from users following recovery from intoxication. J Anal Toxicol. 2012 Nov-Dec;36(9):638-46. doi: 10.1093/jat/bks079. Epub 2012 Oct 7. PMID 23045289
- [Background] Marcotte TD, Heaton RK, Wolfson T, Taylor MJ, Alhassoon O, Arfaa K, Ellis RJ, Grant I. The impact of HIV-related neuropsychological dysfunction on driving behavior. The HNRC Group. J Int Neuropsychol Soc. 1999 Nov;5(7):579-92. doi: 10.1017/s1355617799577011. PMID 10645701
- [Background] Marcotte TD, Rosenthal TJ, Roberts E, Lampinen S, Scott JC, Allen RW, Corey-Bloom J. The contribution of cognition and spasticity to driving performance in multiple sclerosis. Arch Phys Med Rehabil. 2008 Sep;89(9):1753-8. doi: 10.1016/j.apmr.2007.12.049. PMID 18760160
- [Result] Hubbard JA, Hoffman MA, Ellis SE, Sobolesky PM, Smith BE, Suhandynata RT, Sones EG, Sanford SK, Umlauf A, Huestis MA, Grelotti DJ, Grant I, Marcotte TD, Fitzgerald RL. Biomarkers of Recent Cannabis Use in Blood, Oral Fluid and Breath. J Anal Toxicol. 2021 Sep 17;45(8):820-828. doi: 10.1093/jat/bkab080. PMID 34185831
- [Result] Hoffman MA, Hubbard JA, Sobolesky PM, Smith BE, Suhandynata RT, Sanford S, Sones EG, Ellis S, Umlauf A, Huestis MA, Grelotti DJ, Grant I, Marcotte TD, Fitzgerald RL. Blood and Oral Fluid Cannabinoid Profiles of Frequent and Occasional Cannabis Smokers. J Anal Toxicol. 2021 Sep 17;45(8):851-862. doi: 10.1093/jat/bkab078. PMID 34173005
- [Result] Hubbard JA, Smith BE, Sobolesky PM, Kim S, Hoffman MA, Stone J, Huestis MA, Grelotti DJ, Grant I, Marcotte TD, Fitzgerald RL. Validation of a liquid chromatography tandem mass spectrometry (LC-MS/MS) method to detect cannabinoids in whole blood and breath. Clin Chem Lab Med. 2020 Apr 28;58(5):673-681. doi: 10.1515/cclm-2019-0600. PMID 31527291
- [Result] Sobolesky PM, Smith BE, Hubbard JA, Stone J, Marcotte TD, Grelotti DJ, Grant I, Fitzgerald RL. Validation of a liquid chromatography-tandem mass spectrometry method for analyzing cannabinoids in oral fluid. Clin Chim Acta. 2019 Apr;491:30-38. doi: 10.1016/j.cca.2019.01.002. Epub 2019 Jan 4. PMID 30615854
- [Derived] Marcotte TD, Umlauf A, Grelotti DJ, Sones EG, Mastropietro KF, Suhandynata RT, Huestis MA, Grant I, Fitzgerald RL. Evaluation of Field Sobriety Tests for Identifying Drivers Under the Influence of Cannabis: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Sep 1;80(9):914-923. doi: 10.1001/jamapsychiatry.2023.2345. PMID 37531115
- [Derived] Marcotte TD, Umlauf A, Grelotti DJ, Sones EG, Sobolesky PM, Smith BE, Hoffman MA, Hubbard JA, Severson J, Huestis MA, Grant I, Fitzgerald RL. Driving Performance and Cannabis Users' Perception of Safety: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Mar 1;79(3):201-209. doi: 10.1001/jamapsychiatry.2021.4037. PMID 35080588
- See also: Center for Medicinal Cannabis Research, UC San Diego — http://www.cmcr.ucsd.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cannabis: Participants will smoke placebo cannabis with .02% THC ad libitum
- Cannabis With 5.9% THC: Participants will smoke cannabis with 5.9% THC ad libitum
- Cannabis With 13.4% THC: Participants will smoke placebo cannabis with 13.4% THC ad libitum
Period: Overall Study
Arm/Group | Placebo Cannabis | Cannabis With 5.9% THC | Cannabis With 13.4% THC
Started | 65 | 70 | 64
Completed | 63 | 66 | 62
Not Completed | 2 | 4 | 2
Not completed — Oral THC > 5ng/mL prior to treatment (indicating likely recent use) | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Cannabis with .02% THC
- 5.9% THC: Cannabis with 5.9% THC
- 13.4% THC: Cannabis with 13.4% THC
- Total: Total of all reporting groups
Arm/Group | Placebo | 5.9% THC | 13.4% THC | Total
Number analyzed (Participants) | 63 | 66 | 62 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (7.3) | 30.7 (8.8) | 30.9 (8.6) | 29.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 19 | 23 | 73
  Male | 32 | 47 | 39 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8 | 6 | 4 | 18
  Asian | 5 | 8 | 4 | 17
  Hispanic | 15 | 19 | 22 | 56
  Indigenous | 5 | 2 | 1 | 8
  Multiracial | 2 | 3 | 2 | 7
  Non-Hispanic White | 28 | 28 | 27 | 83
  Unknown | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 63 | 66 | 62 | 191

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Drive Score (CDS) From Pre-smoking Simulation
Description: The Composite Drive Score (CDS) is a z-score comprised of key variables from the simulator tasks (SDLP, speed deviation, and task accuracy during the modified Surrogate Reference Task (mSuRT); coherence from the car following task). This outcome reflects the change in CDS from the pre-smoking assessment, at each timepoint.
  The z-score indicates the number of standard deviations away from the mean from the baseline performance for the entire group (n = 191). A Z-score of 0 is equal to the mean of a reference population (in this case the pre-smoking performance for the entire group).
  Higher z-scores at each timepoint indicate worse performance (variables that went in the opposite direction were reflected in order to have all variables have the same direction). When examining the change in Composite Drive Score (this outcome variable), a higher score indicates a decline in performance (e.g., Time 2 minus Time 1).
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Placebo: Placebo Cannabis
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
z-score
  Pre-smoke | -.09 (.64) | .12 (.58) | .01 (.52)
  30 minutes | -.17 (.61) | .46 (.60) | .21 (.60)
  1h 30min | -.13 (.61) | .40 (.66) | .32 (.59)
  3h 30min | -.23 (.59) | .15 (.64) | .04 (.57)
  4h 30min | -.07 (.66) | .09 (.57) | .05 (.59)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p < 0.001, Generalized least squares model

2. Secondary Outcome: Simulator: Standard Deviation of Lateral Position (SDLP)
Description: This measures the standard deviation of lateral (lane) position, or the degree to which the participant "swerves" within the road lane on the driving simulation during the modified Surrogate Reference Task (mSuRT). The range is from .39 to 3.33. A higher score indicates worse performance.
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
z-score
  Pre-smoking | 1.09 (.36) | 1.20 (.36) | 1.11 (0.35)
  30 min | 1.07 (.33) | 1.24 (.36) | 1.19 (.36)
  1h 30min | 1.06 (.31) | 1.31 (.39) | 1.23 (.42)
  3h 30min | 1.10 (.31) | 1.25 (.35) | 1.20 (.42)
  4h 30min | 1.10 (.36) | 1.25 (.37) | 1.18 (.42)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.022, Generalized least squares model; Raw data converted to z-score based on pre-smoking performance of entire sample

3. Secondary Outcome: Simulator: Speed Deviation
Description: The variability in speed during the modified Surrogate Reference Test (mSuRT). The speed is in miles per hour. Range is from .17 to 12.85. A higher score indicates worse performance.
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: miles per hour
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
miles per hour
  Pre-smoking | 2.13 (1.81) | 2.61 (1.97) | 2.63 (1.98)
  30 min | 2.03 (1.31) | 3.04 (1.71) | 2.99 (2.05)
  1h 30min | 2.49 (1.70) | 2.97 (1.93) | 3.01 (2.03)
  3h 30min | 2.15 (1.89) | 3.04 (2.16) | 2.65 (1.72)
  4h 30min | 2.34 (1.82) | 2.92 (2.10) | 2.34 (1.71)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.283, Generalized least squares model

4. Secondary Outcome: Simulator: Correct Hits on mSuRT
Description: The number of times the participant touched the correct stimulus (circle) on the iPad, during modified Surrogate Reference Task (mSuRT). Range is from 8 to 32. A higher score is a better score.
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: count of correct responses
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
count of correct responses
  Pre-smoking | 30.7 (1.80) | 29.9 (2.76) | 30.6 (1.42)
  30 min | 30.9 (1.71) | 28.7 (4.23) | 30.3 (2.54)
  1h 30min | 30.3 (2.16) | 29.6 (2.56) | 30.4 (1.69)
  3h 30min | 30.4 (2.73) | 29.7 (2.61) | 30.7 (1.40)
  4h 30min | 31.0 (1.44) | 30.3 (2.65) | 31.1 (1.05)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.0503, Generalized estimating equations model

5. Secondary Outcome: Simulator: Car Following - Coherence
Description: Coherence is the correlation (0 to 1) between the participant and the lead car (which speeds up and slows down), representing the participant's ability to accurately speed up and slow down similarly to the lead car. Range of scores is from .01 to .97. A higher score is a better score.
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: Correlation coefficient
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
Correlation coefficient
  Pre-smoking | .76 (.19) | .73 (.18) | .76 (.15)
  30 min | .79 (.13) | .66 (.20) | .71 (.17)
  1h 30min | .77 (.16) | .65 (.23) | .68 (.19)
  3h 30min | .80 (.15) | .74 (.18) | .74 (.17)
  4h 30min | .75 (.16) | .74 (.18) | .71 (.17)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.024, Generalized least squares model

6. Secondary Outcome: Simulator: Response Delay - Car Following
Description: Time delay (in seconds) in responding to changes in the lead car's speed. Range is from -5.8 to 6.0. A higher score indicates a worse score.
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
seconds
  Pre-smoking | 2.92 (1.15) | 3.32 (1.23) | 3.58 (1.24)
  30 min | 2.86 (1.05) | 3.44 (1.15) | 3.55 (1.06)
  1h 30min | 2.80 (.99) | 3.25 (1.28) | 3.49 (1.04)
  3h 30min | 2.61 (1.04) | 2.83 (1.05) | 3.23 (1.18)
  4h 30min | 2.93 (1.05) | 3.00 (1.10) | 3.50 (1.17)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.716, Generalized least squares model; The outcome was standardized prior to analyses

7. Secondary Outcome: Simulator: Distance From Lead Car - Car Following
Description: The outcome is distance from the lead car (in virtual feet) during the Car Following Task
Time Frame: Participants are assessed pre-smoking, and then approximately 30m, 1h 30m, 3h 30m and 4h 30m post-smoking
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
feet
  Pre-smoking | 153 (41) | 156 (41) | 163 (35)
  30 min | 143 (36) | 165 (39) | 164 (39)
  1h 30min | 144 (34) | 160 (38) | 165 (36)
  3h 30min | 129 (33) | 137 (37) | 150 (34)
  4h 30min | 138 (34) | 136 (37) | 151 (36)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = 0.005, Generalized least squares model; The outcome was standardized prior to analysis

8. Secondary Outcome: Tablet Assessment: Dual Attention Missed Switches
Description: The participant follows a moving target (square) with her/his finger, and switches to following a new stimulus when it appears in the corner of the screen. Each participant was classified as to whether he/she missed any of these switches during the trial. The outcome is the proportion of participants within each group who missed at least one switch. The range is from 0 to 1. Higher indicates a worse score.
Time Frame: Participants assessed pre-smoking and 1 hour, 2 hours, 4 hours, and 5 hours after smoking
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
Proportion of participants
  Pre-smoking | 0.095 [0.039 to 0.202] | 0.145 [0.073 to 0.263] | 0.167 [0.087 to 0.290]
  1 hour | 0.095 [0.039 to 0.202] | 0.194 [0.108 to 0.317] | 0.183 [0.099 to 0.309]
  2 hours | 0.175 [0.095 to 0.295] | 0.161 [0.084 to 0.281] | 0.233 [0.138 to 0.363]
  4 hours | 0.191 [0.106 to 0.313] | 0.177 [0.096 to 0.299] | 0.167 [0.087 to 0.290]
  5 hours | 0.095 [0.039 to 0.202] | 0.129 [0.061 to 0.244] | 0.183 [0.099 to 0.309]
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = .366, Generalized Estimating Equations model

9. Secondary Outcome: Tablet Assessment: Lane Tracking Standard Deviation
Description: The participant is to rotate the iPad in order to keep a round object in the center, between two lines (lanes). This measure is the standard deviation of the position of the round object during the task (in essence, how much "swerving" there is within the lane). The range is from 8.2 to 189.4. A higher score indicates worse performance.
Time Frame: Participants assessed pre-smoking and 1 hour, 2 hours, 4 hours, and 5 hours after smoking
Measure: Mean (Standard Deviation); unit: standard deviation of position
Groups:
- 5.9% THC; 13.4% THC: Cannabis with 13.4% THC
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
standard deviation of position
  Pre-smoking | 26.9 (9.53) | 30.9 (23.7) | 27.2 (9.67)
  1 hour | 28.7 (13.4) | 30.9 (15.7) | 32.1 (21.7)
  2 hours | 28.4 (10.3) | 27.6 (10.2) | 27.4 (10.4)
  4 hours | 28.1 (13.3) | 29.9 (15.5) | 28.6 (14.8)
  5 hours | 26.4 (10.8) | 25.4 (8.39) | 25.3 (13.8)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = .225, Generalized least squares model; Outcome was log10 transformed prior to analyses

10. Secondary Outcome: Tablet Assessment: Visual Spatial Learning Test Number Correct
Description: Assessment of short-term memory for abstract figures. The participant is to memorize abstract figures and their locations on a 3 x 3 grid. After initial viewing (10 seconds), the figures go away for either 4, 12, or 24 seconds. The participant is then to identify which figures were in the initial viewing (from a list at the bottom of the screen), and place them at the correct location. This is the number of correctly identified figures. The range is from 0 to 12. A higher score indicates better performance.
Time Frame: Participants assessed pre-smoking and 1 hour, 2 hours, 4 hours, and 5 hours after smoking
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
number of correct responses
  Pre-smoking | 9.9 (2.3) | 9.7 (2.7) | 10.1 (2.2)
  1 hour | 9.1 (2.8) | 8.4 (2.6) | 9.3 (2.7)
  2 hours | 8.9 (3.1) | 8.7 (2.6) | 8.9 (2.7)
  4 hours | 8.5 (3.0) | 8.3 (2.9) | 8.8 (2.5)
  5 hours | 9.3 (2.9) | 8.5 (3.0) | 9.5 (3.0)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = .592, Generalized least squares model; The outcome was transformed using logit function prior to analyses. Model included treatment (3 groups), time (5 times), and their interaction

11. Secondary Outcome: Tablet Assessment: Time Estimation
Description: The participant is to estimate the amount of time that has passed while performing a secondary task. This outcome is the ratio of 1) the estimated time that has passed (seconds), divided by 2) the actual amount of time that has passed. The range is from 0.204 to 1.89. A higher score indicates a better performance.
Time Frame: Participants assessed pre-smoking and 1 hour, 2 hours, 4 hours, and 5 hours after smoking
Measure: Mean (Standard Deviation); unit: Ratio of estimated/actual time
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
Ratio of estimated/actual time
  Pre-smoking | 0.75 (0.19) | 0.83 (0.30) | 0.77 (0.22)
  1 hour | 0.79 (0.21) | 0.89 (0.30) | 0.85 (0.24)
  2 hours | 0.83 (0.20) | 0.96 (0.30) | 0.87 (0.27)
  4 hours | 0.85 (0.23) | 0.93 (0.23) | 0.86 (0.21)
  5 hours | 0.83 (0.20) | 0.89 (0.28) | 0.85 (0.21)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = .294, Generalized least squares model

12. Secondary Outcome: Tablet Assessment: Balance
Description: While standing and keeping their feet still, this is a measure of the participant's "sway", which is the total distance that the participant's body moved (in meters) from his/her initial vertical position. This was measured using an accelerometer placed on the participant's back. The range of scores is from .222 to 1.661. A higher score indicates worse performance.
Time Frame: Participants assessed pre-smoking and 1 hour, 2 hours, 4 hours, and 5 hours after smoking
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
meters
  Pre-smoking | 0.358 (0.058) | 0.360 (0.067) | 0.356 (0.058)
  1 hour | 0.342 (0.054) | 0.376 (0.090) | 0.363 (0.129)
  2 hours | 0.351 (0.053) | 0.394 (0.161) | 0.414 (0.254)
  4 hours | 0.354 (0.058) | 0.386 (0.131) | 0.377 (0.133)
  5 hours | 0.368 (0.059) | 0.371 (0.054) | 0.365 (0.072)
Statistical Analysis 1: Comparison: Placebo vs 5.9% THC vs 13.4% THC; Test type: Superiority; p = .144, Generalized least squares model

13. Secondary Outcome: THC Concentrations: Correlation Between Blood and Oral Fluid
Description: Spearman's correlation between THC concentrations in whole blood and oral fluid. Higher scores are better.
Time Frame: Approximately 15 minutes post-smoking
Measure: Number (95% Confidence Interval); unit: Spearman's rho
Groups:
- 5.9% THC: Participants smoking 5.9% THC cannabis
- 13.4% THC: Group smoking 13.4% THC
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
Spearman's rho | 0.217 [-0.034 to 0.443] | 0.414 [0.190 to 0.598] | 0.249 [-0.003 to 0.471]
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Spearman's correlation; p = 0.090, Spearman's correlation
Statistical Analysis 2: Comparison: 5.9% THC; Test type: Other — Spearman's correlation; p = .0006, Spearman's correlation
Statistical Analysis 3: Comparison: 13.4% THC; Test type: Other — Spearman's correlation; p = 0.053, Spearman's correlation

14. Secondary Outcome: THC Concentrations: Correlation Between Whole Blood and Breath
Description: Spearman's correlation between THC concentrations in whole blood and breath
Time Frame: Approximately 15 minutes post-smoking
Measure: Number (95% Confidence Interval); unit: Spearman's rho
Arm/Group | Placebo | 5.9% THC | 13.4% THC
Number analyzed (Participants) | 63 | 66 | 62
Spearman's rho | 0.134 [-0.120 to 0.371] | -0.258 [-0.472 to -0.015] | -0.176 [-0.410 to 0.079]
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Spearman's correlation; p = 0.300, Spearman's correlation
Statistical Analysis 2: Comparison: 5.9% THC; Test type: Other — Spearman's correlation; p = 0.038, Spearman's correlation
Statistical Analysis 3: Comparison: 13.4% THC; Test type: Other — Spearman's correlation; p = 0.175, Spearman's correlation

ADVERSE EVENTS:
Time Frame: One day (acute administration)
Groups:
- Placebo Cannabis: Placebo Cannabis (.02% THC)
- Cannabis With 5.9% THC: Cannabis with 5.9% THC, smoked ad libitum
- Cannabis With 13.4% THC: Cannabis with 13.4% THC, smoked ad libitum
Arm/Group | Placebo Cannabis | Cannabis With 5.9% THC | Cannabis With 13.4% THC
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/70 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/70 | 0/64
Other Adverse Events (participants affected / at risk) | 2/65 | 15/70 | 5/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cannabis (N=65) | Cannabis With 5.9% THC (N=70) | Cannabis With 13.4% THC (N=64)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Sweats (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Blood Pressure Decreased (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Blood Pressure Increased (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Heart Rate Abnormal (Cardiac disorders) | 0 (0) | 12 (12) | 1 (1)
Cervicalgia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fainting (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort in arm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Venous catheter was used to collect blood
Swollen arm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Venous catheter was used to collect blood
Numbness in arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Venous catheter was used to collect blood
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT02849587/Prot_SAP_001.pdf